CLINICAL TRIAL: NCT01476800
Title: A Phase 1, Open-Label, Two-Period, One-Sequence Crossover Study to Assess Pharmacokinetic Interaction of Multiple Dose Ketoconazole on Single Dose YM178 Oral Controlled Absorption System (OCAS) in Healthy Male and Female Adult Volunteers
Brief Title: A Study to Assess Pharmacokinetic Interaction of Multiple Dose Ketoconazole on Single Dose YM178 Oral Controlled Absorption System (OCAS) in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: 178-CL-036
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Healthy Subjects; Pharmacokinetics of YM178
Keywords: Drugs, Investigational; pharmacokinetics; Urinary Bladder, Overactive; YM178; Mirabegron
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- YM178 OCAS alone (Experimental)
  Interventions: Drug: YM178 OCAS
- Ketoconazole alone (Active Comparator)
  Interventions: Drug: Ketoconazole
- YM178 OCAS and ketoconazole (Experimental)
  Interventions: Drug: YM178 OCAS

INTERVENTIONS:
Drug: YM178 OCAS — oral
  Other Names: mirabegron
  Arms: YM178 OCAS alone; YM178 OCAS and ketoconazole
Drug: Ketoconazole — oral
  Other Names: Nizoral
  Arms: Ketoconazole alone

SUMMARY:
The purpose of this study is to assess the pharmacokinetic interaction of multiple-dose ketoconazole on single-dose YM178 OCAS and the safety and tolerability of YM178 OCAS alone and in combination with ketoconazole in healthy adult volunteers.

DETAILED DESCRIPTION:
A single oral dose of YM178 OCAS will be administered on 2 separate occasions: alone on Day 1 of Period 1 and during multiple- dosing of ketoconazole on Day 4 of Period 2. In Period 2, an oral dose of ketoconazole will be administered once daily on Days 1-9.

ELIGIBILITY:
Inclusion Criteria:

* The subject, if female, must be surgically sterile (must be documented), post-menopausal (defined as at least two years without menses), or must be using double-barrier contraception or a non-hormonal IUD
* The subject, if female, must be non-lactating, and have a negative serum pregnancy test result during the study
* The subject must be in good health
* The subject must weigh at least 45 kg, and have a Body Mass Index (BMI) between 18 and 30 kg/m^2, inclusive
* The subject must have normal clinical laboratory test results or, if abnormal, are not clinically significant
* The subject must have a normal 12-lead electrocardiogram (ECG) (including normal interval durations). If abnormal, the interval durations must be deemed not clinically significant and must not exceed the following values: PR intervals must not exceed 220 milliseconds and QTc values must not exceed 450 milliseconds in Males or 470 milliseconds in females
* The subject must have negative drug and alcohol toxicology screens during the study. Any subject who tests positive for drugs or alcohol during the study will be terminated

Exclusion Criteria:

* The subject has a history of clinically significant illness (e.g., cardiovascular, hepatic, renal, or gastrointestinal abnormality within past 3 months that would preclude participation in the study
* The subject is known to have hepatitis or is positive for hepatitis A antibody IgM, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or has a positive result to tests for HIV-1 and/or HIV-2 antibodies
* The subject is known to have hypersensitivity to YM178, or ketoconazole or other imidazole compounds
* The subject has a resting supine pulse <50 bpm or >90 bpm
* The subject has orthostasis (change in pulse rate with orthostatic maneuver of >20 bpm or to a level ≥ 120 bpm)
* The subject is taking any oral hormonal contraceptive
* The subject is taking a potential inhibitor of CYP3A4 or CYP2D6
* The subject has received or is anticipated to receive a prescription systemic or topical medication within past 14 days or any long-active treatments (e.g., depot formulation) within past 30 days
* The subject has received any other-the-counter medication including herbal medicines within past 14 days (occasional use of acetaminophen of up to 2000 mg/day but not more than 4 days per week is permitted)
* The subject is currently participating in another clinical trial and/or is taking or has been taking an investigational drug in the past 30 days (or 10 half-lives of the drug, whichever is longer)
* The subject anticipates an inability to abstain from alcohol, or caffeine use, or from grapefruit and grapefruit juice from 48 hours prior to the administration of the first dose of YM178 on Day 1 of Period 1 and throughout the duration of the study
* The subject has used tobacco-containing products and nicotine or nicotine-containing products in past six months
* The subject consumes more than 5 units of alcoholic beverages (one unit is 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits) per week or has a history of substance abuse, drug addiction, or alcoholism within past 2 years.
* The subject has had any blood donation or significant loss of blood or has received transfusion of any blood or blood products within 56 days of study initiation or has donated plasma within 7 days of study initiation.
* The subject has a history of psychiatric illness within past 10 years or is incapable of being compliant with the study procedures
* The subject is unable to understand verbal and/or written English or any other language in which a certified translation of the informed consent is available
* The subject has a history of benign prostatic hypertrophy or urinary incontinence

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-07; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) variable for YM178: Area under the plasma concentration - time curve from time of dosing to infinity (AUCinf) | Up to Day 7 in Period 1 and up to Day 10 in Perod 2
PK Variable for YM178: Maximum concentration (Cmax) | Up to Day 7 in Period 1 and up to Day 10 in Perod 2

SECONDARY OUTCOMES:
Safety assessed by recording of adverse events, vital signs, laboratory assessments, electrocardiograms (ECGs) and physical exams | Up to Day 7 in Period 1 and up to Day 10 in Period 2

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- MDS Pharma Services (US) Inc., Lincoln, Nebraska, United States